CLINICAL TRIAL: NCT05725473
Title: Clinical Efficacy and Safety of Endoscopic Dilatation With Eso-Filp in Benign Esophageal Strictures
Acronym: ESO-FLIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3022
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eso-Flip (Experimental): Dilatation with Eso-Flip
  Interventions: Device: Eso-Flip

INTERVENTIONS:
Device: Eso-Flip — Dilatation with Eso-FLIP

SUMMARY:
Benign esophageal strictures are frequently seen in endoscopic practice and are caused by a variety of esophageal disorders, including peptic, radiotherapy-induced and caustic injuries, Schatzki ring, eosinophilic esophagitis (EoE), and strictures after surgical resection (anastomotic) or endoscopic resection (endoscopic mucosal resection-EMR- and endoscopic submucosal dissection-ESD), and ablative therapies (Radiofrequency, Cryotherapy and Argon-plasma coagulation).

Endoscopic dilation is the first treatment step for benign esophageal strictures. Two types of dilators are available, namely, through-the-scope balloon dilators, with or without a guidewire, and wire-guided bougie dilators. Bougie dilators are used for simple strictures and for strictures in the proximal esophagus, especially anastomotic strictures. Bougie dilators exert a combined radial and longitudinal force, which may increase the risk of perforation. Bougie dilators allow, however, sensing the degree of resistance during dilation, and thereby help determining increasing bougie sizes during next-step dilations. Through the-scope balloon dilators are preferred for complex strictures. Balloons dilators allow direct visualization and control of the radially applied dilation force. In literature, both dilation techniques appear to be equally effective and safe in the management of esophageal strictures, showing no differences in terms of risks of AEs About 30 years ago, the "rule of three" has been published. This rule dictated the extent of dilation during any endoscopic session (i.e., no more than three dilators successively larger than the first dilator to meet resistance were passed) and has been used by endoscopists to reduce the risk of perforation. However, the safety of the "rule of three" has never been demonstrated. Moreover, a recent study suggests that more than three dilation steps per session may be considered for esophageal strictures, with the exception of malignant strictures. The EsoFLIP (Medtronic Inc., Shoreview, MN, USA) is a novel dilation balloon that provides real-time, objective visualization and monitoring of therapeutic dilation. EsoFLIP utilizes high-resolution impedance planimetry to provide real-time measurements (diameter and cross-sectional area) of the stenotic area before, during, and at the end of the dilation without the need of fluoroscopy.

In 2013, technical feasibility and safety of the EsoFLIP in esophago-gastric junction (EGJ) dilation have been demonstrated on porcine models. In a small first pilot study, the technical feasibility of the EsoFLIP device in 10 patients with achalasia has been demonstrated. A second study reported short-term efficacy, both objective (improvement in barium column) and subjective (improvement in Eckardt score), in 28 patients managed using the FLIP hydraulic balloon dilator. Very limited data are currently available in the literature on the use of EsoFLIP in benign esophageal strictures dilation. Potential advantages of the use of EsoFLIP are dilation without fluoroscopy and associated radiation, control of dilation sizes to generate the desired dilation effect and assessment of stricture size and the response to dilatation immediately following dilation.

In a small single centre retrospective study on 19 paediatric patients, use of EsoFLIP hydraulic dilation was safe and provided a larger diameter increase compared with standard balloon dilation, but this was not statistically significant likely because of the small cohort size. The study also suggested that procedure time and fluoroscopy time were shorter in the EsoFLIP cases when compared to other traditional dilation methods. Esophageal dilation using EsoFLIP may yield a larger diameter change increasing the interval between a dilatation procedure and the following one and may potentially reduce procedure time when compared to traditional balloon dilation.

There is currently no published prospective study about dilation with EsoFLIP in adult patients affected by benign esophageal strictures. The endoluminal functional lumen imaging probe, EndoFLIP™ (Medtronic, Minneapolis, MN, USA) (FLIP), is a tool that utilizes impedance planimetry, a technique for performing balloon distention in the alimentary track, to obtain dynamic measurements of any sphincters including the diameter, cross-sectional area (CSA), and distensibility index (DI). Diseases where Endo-FLIP has been employed include esophageal stenosis, reflux esophagitis, eosinophilic esophagitis, gastroparesis, anal sphincter disease, achalasia, and it has also been used in peroral endoscopic myotomy.

ELIGIBILITY:
Inclusion Criteria:

* Dysphagia due to benign esophageal stricture (e.g. surgery, radiation therapy, caustic ingestion, peptic injury, photodynamic therapy, EoE)
* A benign esophageal stricture requiring endoscopic esophageal dilation (naïve and refractory to previous treatments)

Exclusion Criteria:

* Patient with known esophageal motility disorder (such as achalasia)
* Age < 18 years at moment of inclusion in retrospective cohort study
* Patient unable to give consent to the participation of the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | 12 months
  Reduction of severity and frequency of dysphagia (Brief Esophageal Dysphagia Questionnaire, Likert scale, BEDQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No